CLINICAL TRIAL: NCT05193448
Title: A Non-interventional Ambispective Real-world Cohort of rEfractory and reLapsed FLT3 Mutated Acute MyEloid Leukemia Patients Treated With Gilteritinib in FrANCE
Brief Title: A Non-interventional Ambispective Real-world Cohort of rEfractory and reLapsed (R/R) FLT3 Mutated Acute MyEloid Leukemia (AML) Patients Treated With Gilteritinib in FrANCE
Acronym: ELEGANCE
Status: Completed | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Other Study IDs: ELEGANCE
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Refractory AML; Relapsed Adult AML; FLT3-TKD Mutation; FLT3-ITD
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gilteritinib is available in early access in France through Temporary Authorisation of Use (or ATU program) since March 2019. The ATU program reflects a real-life treatment situation and the related clinical data would help to better understand the benefit/risk profile of gilteritinib and to better document gilteritinib efficacy and safety in patients who received midostaurine in First Line (1L) setting.

The main objective is to describe gilteritinib effectiveness in FLT3 (Fms Related Tyrosine Kinase 3) -mutated AML patients in Refractory/Relapsed(R/R) situation treated in the context of early access program to gilteritinib in France through Temporary Authorisation of Use, the so-called ATU program, and the post ATU period from marketing authorisation to launch when reimbursement and price are published.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years at AML diagnosis
* Patients that started gilteritinib during ATU and post-ATU period from 19th March 2019 to 30th March2021
* Patients diagnosed with refractory or relapsed AML as defined by the World Health Organization (WHO) Classification
* Patients with FLT3 genetic testing performed at diagnosis and/or at R/R (if available)
* Gilteritinib with or without other drug (chemotherapy, hypomethylating agent, hydroxyurea, etc.)

Exclusion Criteria:

* Newly diagnosed AML patients
* Participant opposed to the collection and analysis of their medical data
* Prescription of gilteritinib out of the scope of its marketing authorisation approval such as post HSCT maintenance in patients in first complete remission after intensive chemotherapy
* persons placed in curatorship,guardianship or guardianship orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥18 years of age FLT3-mutated R/R AML as defined by the WHO Classification between the periods of March 1st, 2019 to September 30, 2021 allowing 6-months follow-up for the last patient included (March, 19 2019 to September 18, 2019 for French "ATU nominative"; September 18, 2019 to January 08, 2020 for French "ATU de cohorte"; January 08, 2020 to March 30, 2021 for "post ATU" period) treated in virtually all AML center in France
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Gilteritinib effectiveness in FLT3-mutated AML patients in R/R situation | 6 months
  best response obtained according to European Leukemia Net (ELN) 2017 recommendations and ADMIRAL definitions effectiveness will also described in the following subgroups : refractory after 1st line chemo, 1rst relapse =< 6 months after Complete Remission (CR) 1, 1st relapse > 6 months after CR1, refractory after 1 st relapse salvage treatment, beyond the first relapse (>= 2nd relapse), post Hematopoietic Stem Cell Transplantation (HSCT), post 1L midostaurine and by ELN 2017 risk groups

CONTACTS AND LOCATIONS:
Locations (38):
- France (38):
  - Amiens CHU, Amiens
  - Angers CHU, Angers
  - Avignon CH, Avignon
  - Bayonne CH, Bayonne
  - Besançon CHU, Besançon
  - Brest CHU, Brest
  - Caen CHU, Caen
  - CERGY PONTOISE - CH René Dubos, Cergy-Pontoise
  - CHU Estaing, Clermont-Ferrand
  - Corbeil-Essonnes - Ch Sud Francilien, Corbeil-Essonnes
  - Créteil CHU HENRI MONDOR, Créteil
  - Dijon CHU, Dijon
  - Grenoble CHU, Grenoble
  - Le Mans CH, Le Mans
  - Limoges CHU, Limoges
  - Lyon sud CHU, Lyon
  - Marseille IPC, Marseille
  - Meaux CH de l'Est francilien, Meaux
  - METZ-THIONVILLE CHR- Hôpital de Mercy, Metz
  - Montpellier - Chu Saint Eloi, Montpellier
  - Nantes CHU, Nantes
  - Nice CHU, Nice
  - Nimes CHU, Nîmes
  - Paris La Pitié salpetrière, Paris
  - Paris Necker, Paris
  - Paris Saint Louis, Paris
  - Bordeaux CHU, Pessac
  - Reims CHU, Reims
  - Rennes CHU, Rennes
  - roubaix CH, Roubaix
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Saint Quentin CH, Saint-Quentin
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - Tours CHU, Tours
  - Troyes CH, Troyes
  - Nancy CHU, Vandœuvre-lès-Nancy
  - Versailles CH, Versailles
  - Villejuif IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No